CLINICAL TRIAL: NCT07220616
Title: A Phase 1/2, Multicenter, Open-Label, Multi-Cohort, First-in Human Trial of DS3790a, for Hematological Malignancies
Brief Title: A First-in-Human Trial of DS3790a in Participants With Hematological Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS3790-076; 2025-522595-87-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-21; First posted 2025-10-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hematological Malignancies
Keywords: Hematological Malignancies; DS3790a
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Drug Combinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Monotherapy Dose Escalation Phase (Experimental): Participants with hematological malignancies who received DS3790a monotherapy.
  Interventions: Drug: DS3790a
- Monotherapy Dose Expansion Phase (Experimental): Participants with hematological malignancies who received DS3790a monotherapy.
  Interventions: Drug: DS3790a
- Cohort A Combination Dose-escalation Phase (Experimental): Participants with hematological malignancies who received DS3790a monotherapy and selected combination regimen.
  Interventions: Drug: DS3790a; Drug: Combination drug
- Cohort A Randomization/Optimization Phase (Experimental): Participants with hematological malignancies who received DS3790a monotherapy and selected combination regimen.
  Interventions: Drug: DS3790a; Drug: Combination drug
- Cohort A Phase 2 (Experimental): Participants with hematological malignancies who received DS3790a monotherapy and selected combination regimen.
  Interventions: Drug: DS3790a; Drug: Combination drug
- Cohort B Combination Dose-escalation Phase (Experimental): Participants with hematological malignancies who received DS3790a monotherapy and selected combination regimen.
  Interventions: Drug: DS3790a; Drug: Combination drug
- Cohort B Randomization/Optimization Phase (Experimental): Participants with hematological malignancies who received DS3790a monotherapy and selected combination regimen.
  Interventions: Drug: DS3790a; Drug: Combination drug
- Standard of Care (Active Comparator): Participants with hematological malignancies who received standard of care (SoC).
  Interventions: Drug: Combination drug

INTERVENTIONS:
Drug: DS3790a — Administered as specified in the protocol
  Arms: Cohort A Combination Dose-escalation Phase; Cohort A Phase 2; Cohort A Randomization/Optimization Phase; Cohort B Combination Dose-escalation Phase; Cohort B Randomization/Optimization Phase; Monotherapy Dose Escalation Phase; Monotherapy Dose Expansion Phase
Drug: Combination drug — Administered as specified in the protocol
  Arms: Cohort A Combination Dose-escalation Phase; Cohort A Phase 2; Cohort A Randomization/Optimization Phase
Drug: Combination drug — Administered as specified in the protocol
  Arms: Cohort B Combination Dose-escalation Phase; Cohort B Randomization/Optimization Phase; Standard of Care

SUMMARY:
This clinical trial is designed to assess the safety, preliminary efficacy, and pharmacokinetics (PK) of DS3790a monotherapy and combination regimens in participants with hematological malignancies.

DETAILED DESCRIPTION:
DS3790a may be effective in the treatment of patients with hematological malignancies. The primary objective of this study will assess the safety and preliminary efficacy of DS3790a monotherapy and combination regimens.

ELIGIBILITY:
To be eligible to participate in this trial, an individual must meet all the following criteria:

1. Sign and date the ICF, prior to the start of any trial-specific procedures.
2. Adults ≥18 years at the time the ICF is signed
3. History of one of the histologically documented hematologic malignancies according to the 5th edition of WHO classification as specified in the protocol.
4. Agree to provide tumor samples as specified in the protocol.
5. ECOG PS of 0, 1 or 2 assessed no more than 14 days prior to initiation of trial intervention.
6. Has adequate organ and bone marrow function as assessed by local laboratory within 14 days prior to initiation of trial intervention as specified in the protocol.
7. Has an LVEF ≥50% by either an ECHO or MUGA within 28 days before the trial starts.
8. Life expectancy of at least 3 months.
9. Is willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other trial procedures, and trial restrictions.
10. A woman of childbearing potential is eligible to participate if she meets all criteria as specified in the protocol.
11. A male participant capable of producing sperm is eligible to participate if he agrees to all criteria as specified in the protocol.

An individual who meets any of the following criteria will be excluded from participating in this trial:

1. Prior Allo-SCT.
2. Prior solid organ transplantation.
3. Inadequate washout period before initiation of trial intervention as specified in the protocol
4. Evidence of brain or leptomeningeal disease (spinal cord or CNS metastases) based on history and physical examination, unless treated and with radiologically documented lack of progression within 4 weeks prior to initiation of trial intervention.
5. Uncontrolled or significant cardiovascular disease as specified in the protocol.
6. Any of the following within the past 6 months prior to enrollment: cerebrovascular accident, transient ischemic attack, or other arterial thromboembolic event.
7. Has a history of (noninfectious) ILD/pneumonitis that required corticosteroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
8. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
9. Has been diagnosed with another malignancy within the previous 3 years
10. Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE Version 5.0, Grade ≤1 or baseline.
11. Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection.
12. Has active or uncontrolled HBV, HCV, or HIV infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting Dose-limiting Toxicities, Treatment-emergent Adverse Events, Serious Adverse Events, Adverse Events of Special Interest, and Deaths in Participants With Hematological Malignancies | Baseline up to 5 years
  Adverse events (AEs) will be graded using NCI-CTCAE version 5.0.
Complete Response in Participants With Hematological Malignancies by Blinded Independent Central Review (Cohort A Randomization Optimization Phase, Cohort A Phase 2) | Baseline up to 5 years
  Complete Response (CR) is defined as participants with CR as measured by BICR assessment.
Complete Response in Participants With Hematological Malignancies by Investigator Assessment (Cohort B Randomization Optimization Phase) | Baseline up to 5 years
  Complete Response (CR) is defined as participants with CR as measured by investigator assessment.

SECONDARY OUTCOMES:
Objective Response by Investigator Assessment In Participants With Hematological Malignancies | Baseline up to 5 years
  Objective response (OR) is defined as participants with complete response (CR) or partial response (PR) as measured by investigator assessment.
Complete Response in Participants With Hematological Malignancies by Investigator Assessment (Monotherapy Dose Escalation, Cohort A Combination Dose Escalation, Cohort B Combination Dose Escalation) | Baseline up to 5 years
  Complete response (CR) is defined as participants with CR as best overall response (BOR) as measured by investigator assessment.
Disease Control in Participants With Hematological Malignancies by Investigator Assessment (Monotherapy Dose Escalation, Cohort A Combination Dose Escalation, Cohort B Combination Dose Escalation) | Baseline up to 5 years
  Disease control (DC) is defined as participants with CR, PR or stable disease as BOR as measured by investigator assessment.
Duration of Complete Response and Duration of Response in Participants With Hematological Malignancies by Investigator Assessment (Monotherapy Dose Escalation, Cohort A Combination Dose Escalation, Cohort B Combination Dose Escalation) | Baseline up to 5 years
  Duration of Complete Response (DoCR) is defined as the time from the date of first documentation of CR to the first documentation of objective tumor progression by investigator assessment or to death due to any cause, whichever occurs first. DoCR will be calculated for responders (CR) only.
  Duration of Response (DoR) is defined as the time from the date of first documentation of objective response (CR or PR) to the first documentation of objective tumor progression by investigator assessment or to death due to any cause, whichever occurs first. DoR will be calculated for responders (CR or PR) only.
Time to Response in Participants With Hematological Malignancies by Investigator Assessment (Monotherapy Dose Escalation, Cohort A Combination Dose Escalation, Cohort B Combination Dose Escalation) | Baseline up to 5 years
  Time to Response (TTR) is defined as the time from the date of the start of trial intervention or randomization if randomized, to the date of the first documentation of objective response (CR or PR) by investigator assessment. TTR will be calculated for responders (CR or PR) only.
Progression-free Survival Participants With Hematological Malignancies by Investigator Assessment (Monotherapy Dose Escalation, Cohort A Combination Dose Escalation, Cohort B Combination Dose Escalation) | Baseline up to 5 years
  Progression-free Survival (PFS) is defined as time from the date of the start of trial intervention or randomization if randomized, to the date of radiographic disease progression, defined as the first documented objective PD by investigator assessment or death due to any cause.
Overall Survival Participants With Hematological Malignancies by Investigator Assessment (Monotherapy Dose Escalation, Cohort A Combination Dose Escalation, Cohort B Combination Dose Escalation) | Baseline up to 5 years
  Overall Survival (OS) is defined as the time from the date of the start of trial intervention or randomization if randomized, to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that have reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/